CLINICAL TRIAL: NCT06145113
Title: The Effect of Continuous Positive Pressure Ventilation on Symptoms of Acute Mountain Sickness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: Himalayan Rescue Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-2158
Record Dates: First submitted 2023-11-14; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Acute Mountain Sickness
Keywords: Acute mountain sickness; Altitude; CPAP; Positive airway pressure
MeSH Terms: conditions — Altitude Sickness | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant
Masking Description: Each participant will not be aware of which arm to which they have been assigned. The on-site investigator will be responsible for randomization, so they will not be able to be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continuous Positive Airway Pressure - 10cmH2O (Active Comparator): This arm will consist of positive airway pressure at an FiO2 of 21% (ambient air), supplied by CPAP device set to 10cmH2O of pressure, for a total of 2 hours.
  Interventions: Device: Continuous positive airway pressure (CPAP), ResMed AirMini
- Placebo Continuous Positive Airway Pressure - 1cmH2O (Placebo Comparator): This arm will consist of positive airway pressure at an FiO2 of 21% (ambient air), supplied by CPAP device set to 1cmH2O of pressure, for a total of 2 hours. This 1cmH2O is necessary to maintain blinding and will provide minimal therapeutic effect.
  Interventions: Device: Continuous positive airway pressure (CPAP), ResMed AirMini
- Continuous Positive Airway Pressure - 10cmH2O, with supplemental oxygen (Other): This arm will only be enrolled into once the other two arms have been completed. Additional subjects will receive CPAP at 10cmH2O with in-line oxygen (estimated 2-4 liters per minute). This is done to determine if adding supplemental oxygen can further improve symptoms.
  Interventions: Device: Continuous positive airway pressure (CPAP), ResMed AirMini

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP), ResMed AirMini — Consumer CPAP device, designed for use without medical supervision by patients with obstructive sleep apnea. This device is safely used by unconscious patients for several hours at a time. This will be supplied by face mask to awake patients under direct medical supervision.

SUMMARY:
Acute Mountain Sickness (AMS) is a common condition affecting individuals traveling to elevations greater than 2500 meters (8200 feet). While more gradual ascent profiles, as well as the use of acetazolamide, have been shown to decrease the incidence of AMS, it remains a common condition that can affect anyone who travels to altitude. Many pharmacologic options for treatment of AMS exist, however these are not always effective or able to be taken by all patients. Continuous positive airway pressure (CPAP) has been shown in some small studies and reports to be a potential non-pharmacologic method of both preventing and treating AMS. No large trials to validate the efficacy of CPAP in altitude related illness have been done. This study aims to evaluate the degree to which CPAP can improve symptoms of AMS, as well as improve oxygen saturation among individuals traveling in a high altitude location.

DETAILED DESCRIPTION:
AMS is commonly experienced among travelers in all high altitude locations, and can affect anyone who travels to one of these places. This illness can be prevented, and after its symptoms have been started, can be treated with medication, as well as by descending to a lower elevation. The medications for AMS symptoms, including acetazolamide, dexamethasone, and ibuprofen are not always effective, and even when they are, often take considerable time to show their effect. Additionally, not all patients can take these medications. When these medications are not effective, or there is a contraindication to their use, descent to a lower elevation is necessary, however this is not always possible due to weather, debilitating symptoms, or coinciding diagnoses of high altitude pulmonary edema (HAPE) or high altitude cerebral edema (HACE). These situations require a difficult and complicated evacuation, requiring multiple rescuers and heavy equipment, or increased risk of clinical deterioration.

CPAP has been shown to be a potential non-pharmacologic method of both preventing and treating AMS. These limited studies quantified symptoms using the Lake Louise score {LLS}, a clinical tool used to assess the severity of AMS. They showed that LLS among subjects receiving CPAP, LLS lower when using it prophylactically or after AMS symptoms had started, however these were not compared against placebo. Additionally, over the last five years, CPAP devices have become quite portable and battery powered, making them much more suitable for travel to wilderness and high altitude locations. They are also available to consumers at low cost, are designed for travel and weigh less than 1 kg. Taking advantage of these devices' portability, a potential new treatment modality for AMS and other altitude related illnesses exists. Additionally, these devices can offer new solutions for mountain rescue and evacuation of patients suffering from altitude related illness, as these devices have been shown in a yet-to-be-published study to improve oxygen saturation and work of breathing while ambulating and self-carrying the device. Improvements in these assessments has been rapid (less than 2 minutes), potentially offering a more rapid treatment of AMS than existing pharmacologic agents as well. This study will be done in Pheriche, Nepal, as it is a location that has a uniquely elevated prevalence of altitude-related illness.

ELIGIBILITY:
Inclusion Criteria:

* present in Pheriche, Nepal;
* Lake Louise score > 1 (with or without formal AMS diagnosis)

Exclusion Criteria:

* History of chronic respiratory conditions (uncontrolled asthma, COPD, ILD)
* obstructive sleep apnea (if currently using nighttime CPAP)
* congestive heart failure
* coronary artery disease
* history of myocardial infarction
* neurologic disorder
* cognitive disorder
* altered mental status
* pregnancy
* current use of supplemental oxygen
* excessive facial hair,
* claustrophobia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-08-10 (Estimated)

PRIMARY OUTCOMES:
Lake Louise score for symptoms of acute mountain sickness | Prior to intervention, immediately following intervention, morning following intervention
  This is a validated set of criteria used for research purposes to quantify symptoms of acute mountain sickness.
  A Lake Louise score greater than or equal to 3 is considered diagnostic of acute mountain sickness, and ranges from 0 to 15.
  Higher Lake Louise scores are associated with more severe symptoms and level of disability.
  The criteria are as follows:
  Headache: 0-3 Gastrointestinal symptoms: 0-3 Fatigue and/or weakness: 0-3 Dizziness/light-headedness: 0-3 AMS Clinical Functional Score: 0-3

SECONDARY OUTCOMES:
Pulse oximetry | Prior to intervention, continuously while receiving intervention, immediately following intervention, morning following intervention
  Level of peripheral oxygen saturation as measured by pulse oximeter (0-100%)
Heart rate | Prior to intervention, continuously while receiving intervention, immediately following intervention, morning following intervention
  Measured by palpation of peripheral pulses or pulse oximeter (beats per minute)
Respiratory rate | Prior to intervention, continuously while receiving intervention, immediately following intervention, morning following intervention
  Measured by observation of chest rise and fall (breaths per minute)

CONTACTS AND LOCATIONS:
Locations (1):
- Himalayan Rescue Association, Pheriche, Nepal

IPD SHARING:
Plan to Share IPD: Undecided